CLINICAL TRIAL: NCT01250158
Title: First In-vivo Trial of the Liver Percutaneous Isolated Localized Perfusion (PILP) Set for the Treatment of Liver Metastases
Brief Title: Liver-PILP First-in-Man
Acronym: PILP FiM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Device Works NV SA (Industry)
Collaborators: Celerion (Industry); Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CIP 000369
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Liver Metastases
Keywords: Liver Percutaneous Isolated Localized Perfusion; PILP; Isolated Hepatic Perfusion; IHP; Liver metastases; Unresectable liver metastases of different etiologies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liver-PILP kit (Experimental): Liver-PILP kit
  Interventions: Device: Liver-PILP kit

INTERVENTIONS:
Device: Liver-PILP kit — Device: Liver-PILP kit The Liver-PILP kit (three devices) is composed of percutaneous, disposable (single-use), catheter-based devices for targeted, isolated, organ specific (liver), drug delivery and perfusion with high dose drugs.
  1. The Portal Vein Device (PVD): balloon catheter to occlude the portal vein and allow aspiration through a central lumen for portal veno-venous bypass.
  2. The Hepatic Artery Device (HAD): balloon catheter to occlude arterial flow to the liver.
  3. The Vena Cava Device (VCD): catheter based device to isolate and access hepatic outflow to vena cava by creating a closed chamber in vena cava at ostia of the hepatic veins while maintaining central vena cava blood flow from lower extremities to right atrium through reduced central lumen.

SUMMARY:
The purpose of this study is to determine whether the PILP-kit can be safely used, within specific performance parameters, to isolate and perfuse the liver with a chemotherapeutic drug for the treatment of patients with unresectable liver metastases.

DETAILED DESCRIPTION:
The objective of this Medical Device Study, is to demonstrate the feasibility of the liver PILP intervention.

The liver PILP intervention will be considered feasible if the procedure is demonstrated to be safe and the liver PILP kit performs according to specifications.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ECOG (Eastern Cooperative Oncology Group) stages 0 or 1
2. Unresectable metastatic disease predominant in the liver

Exclusion Criteria:

1. More than 60 % tumor involved liver tissue
2. Abnormal vascular anatomy
3. Severe atherosclerosis
4. Dissection and/or thrombotic occlusion and/or aneurysm of the aorta, iliac or hepatic arteries
5. Short suprahepatic vena cava segment (< 1.5 cm)
6. One or both jugular veins are occluded
7. Other severe, concomitant diseases regarding the subject status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the feasibility of the liver PILP intervention. | During intervention and up to 30 days post intervention
  The liver PILP intervention will be considered feasible if the intervention is demonstrated to be safe and the PILP kit performs according to specifications related to localization, flow rates and retrieval of devices.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, Prof MD PhD, Principal Investigator — University Hospitals Leuven, Catholic University; Karen Geboes, Prof MD Phd, Principal Investigator — University Hospital, Ghent; Luc Defreyne, Prof MD PhD, Principal Investigator — University Hospital, Ghent; Marc Van den Eynde, MD, Principal Investigator — University Hospital Louvain Saint-Luc
Locations (3):
- Belgium (3):
  - University Hospital Louvain Saint-Luc, Brussels
  - University Hospital Ghent, Ghent
  - University Hospitals Leuven, Catholic University, Leuven

REFERENCES:
- [Background] Maleux G, Monbaliu D, Verslype C, Casteleyn C, Van De Velde M, Cornillie P, Hoogeveen Y, Van Cutsem E. Percutaneous isolated liver perfusion with occlusion balloons and a catheter-based stent-graft-like perfusion device: an experimental study in a porcine model. Eur Radiol. 2010 Oct;20(10):2372-80. doi: 10.1007/s00330-010-1816-5. Epub 2010 May 22. PMID 20495978